CLINICAL TRIAL: NCT00428701
Title: An Open-Label, Exploratory Trial to Assess Gastric Acid Control in Critically Ill Subjects Receiving Nexium I.V. (Esomeprazole Sodium) 40mg BID for up to 72 Hours
Brief Title: An Open-label, Exploratory Trial to Assess Gastric Acid Control in Critically Ill Subjects Receiving Nexium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00107; Nexium IV ICU Study 107
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gastric Ulcer
Keywords: stress ulcer; critically ill; gastric acid; gastric aspirates; esomeprazole
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Critical Illness | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole Sodium

SUMMARY:
This study is being done to see if Nexium I.V. can reduce and control stomach acid in mechanically ventilated, critically ill patients in an Intensive Care Unit setting.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill male or female subjects 18 years or older who have a baseline gastric aspirate pH less then or equal to 4
* Subjects admitted to an ICU requiring mechanically ventilated
* Subjects will have at least one additional stress ulcer risk factor

Exclusion Criteria:

* Anticipated use of pre-pyloric enteral feeding after screening until the end of study
* Physician estimated survival of less then 96 hours
* Anticipation of major surgery within 96 hours of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to assess gastric acid suppression by esomeprazole iv in critically ill subjects

SECONDARY OUTCOMES:
The secondary objective is to assess time to stable pH greater then or equal to 4 from start of drug

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca
Locations (5):
- United States (5):
  - Research SIte, Newark, Delaware
  - Research Site, Shreveport, Louisiana
  - Research Site, Hershey, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee

REFERENCES:
- [Derived] Metz DC, Fulda GJ, Olsen KM, Monyak JT, Simonson SG, Sostek MB. Intravenous esomeprazole pharmacodynamics in critically ill patients. Curr Med Res Opin. 2010 May;26(5):1141-8. doi: 10.1185/03007991003694308. PMID 20230209